CLINICAL TRIAL: NCT01357733
Title: Early Interim Chemotherapy Response Evaluation by F-18 FDG PET/CT in Diffuse Large B Cell Lymphoma
Brief Title: Interim FDG PET/CT in Diffuse Large B Cell Lymphoma (DLBCL) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Sung Hoon Kim, Chairman of Department of Radiology, The Catholic University of Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KC11EISI0293
Record Dates: First submitted 2011-05-13; First posted 2011-05-23 (Estimated); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: Diffuse, Large B-Cell, Lymphoma; 18F Fluorodeoxyglucose; Radionuclide-Emission Computed Tomography
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interim FDG PET/CT (Other): Single arm study with diagnostic imaging study as the intervention.
  Interventions: Other: Early interim FDG PET/CT after 1 cycle of R-CHOP

INTERVENTIONS:
Other: Early interim FDG PET/CT after 1 cycle of R-CHOP — FDG PET/CT imaging study obtained after 1 cycle of R-CHOP and before the second cycle of R-CHOP

SUMMARY:
Newly diagnosed diffuse large B cell lymphoma (DLBCL) patients who enter this study will receive baseline fluorodeoxyglucose (FDG) positron emission tomography (PET) computed tomography (CT) scan at the time of initial staging. The patients will be diagnosed and undergo initial staging according to The Catholic University Lymphoma Group (CULG) Protocol.

After 1 cycle of rituximab plus cyclophosphamide, doxorubicin, vincristine, prednisone (R-CHOP) chemotherapy, early interim FDG PET/CT will be obtained after the patient recovers from nadir (usually 13 to 16 days after) following the administration of first cycle of R-CHOP,immediately before the second cycle of R-CHOP. The result of early interim FDG PET/CT study will not impact patient management, except in rare case where newly developed lesion is found and biopsy confirmed.

The same PET/CT system and analysis software will be used for all scans from baseline to surveillance for all patients enrolled in this study.

After 3 cycles of R-CHOP, a mid-therapy interim FDG PET/CT will be obtained. Patients with newly developed lesion will receive different chemotherapy regimen, while patients with stable disease, partial metabolic response or complete metabolic response will continue to receive 3 more cycles of R-CHOP.

After the completion of 6 cycles of R-CHOP, the patients will receive a FDG PET/CT scan for response assessment. Selected patients with persistent disease or very bulky tumor volume on initial staging images will receive additional radiation therapy.

The patients will be followed up every 3 months for 2 years from beginning of therapy. Physical examination and lab studies will be done usually every 3 months. Imaging studies will be performed every 3 months alternating between enhanced CT and FDG PET/CT and noted when different schedule is applied for surveillance.

The end points are changes in FDG uptake measurements between the baseline and early interim FDG PET/CT, and between baseline and mid-therapy interim FDG PET/CT scans; response assessment following completion of 6 cycles of R-CHOP with or without radiation therapy assessed by International Workshop Criteria (IWC)+PET and PET Response Criteria in Solid Tumors (PERCIST) guideline; and the 2 year disease free survival.

ELIGIBILITY:
Inclusion Criteria:

* CD20+ diffuse large B cell lymphoma confirmed
* Therapy naïve for lymphoma
* 19 years or older
* Written informed consent

Exclusion Criteria:

* Cannot understand informed consent
* Age under 19 years old
* Previous chemotherapy or radiation therapy for lymphoma
* Known pregnancy or urine/serum hCG (+)
* Unable to lie down still on back for about 30 minutes

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-03-02 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in summed peak standardized uptake value lean (SULpeak) after 3 cycles | baseline and 3 cycles after starting chemotherapy, approximately 49 to 57 days after beginning R-CHOP
  Change in summed SULpeak between baseline FDG PET/CT before chemotherapy and mid-therapy interim FDG PET/CT after 3 cycles in DLBCL patients
Change from baseline in summed SULpeak after 1 cycle | baseline and 1 cycle after starting chemotherapy, approximately 13 to 16 days after beginning R-CHOP
  Change in summed SULpeak between baseline FDG PET/CT before chemotherapy and early interim FDG PET/CT after 1 cycle of R-CHOP in DLBCL patients

SECONDARY OUTCOMES:
2 year disease free survival | up to 2 years after initial diagnosis
  Patients considered to have 2 year disease free survival will be those with complete response after 6 cycles of R-CHOP or isolated persistent disease treated by radiation therapy, AND continuous disease free state for 2 years from the start of therapy (reference standard "success"). All other patients will be considered to not have achieved 2 year disease free survival.
Qualitative response | after chemotherapy with or without radiation therapy is finished, approximately 120 to 210 days after beginning R-CHOP
  Response according to Lugano Classification and Deauville 5 point score. Response according to IWC+PET criteria with qualitative visual analysis of FDG PET/CT using mediastinum as the background reference.
Quantitative response | after chemotherapy with or without radiation therapy is finished, approximately 120 to 210 days after beginning R-CHOP
  Response according to PERCIST criteria with change in summed SULpeak in the FDG PET/CT as the background reference.

CONTACTS AND LOCATIONS:
Overall Officials: Seok-Goo Cho, MD, PhD, Principal Investigator — The Catholic University of Korea; Joo Hyun O, MD, Principal Investigator — The Catholic University of Korea
Locations (1):
- The Catholic University of Korea Seoul St. Mary's Hospital, Seoul, South Korea

REFERENCES:
- [Background] Wahl RL, Jacene H, Kasamon Y, Lodge MA. From RECIST to PERCIST: Evolving Considerations for PET response criteria in solid tumors. J Nucl Med. 2009 May;50 Suppl 1(Suppl 1):122S-50S. doi: 10.2967/jnumed.108.057307. PMID 19403881
- [Background] Michallet AS, Trotman J, Tychyj-Pinel C. Role of early PET in the management of diffuse large B-cell lymphoma. Curr Opin Oncol. 2010 Sep;22(5):414-8. doi: 10.1097/CCO.0b013e32833d5905. PMID 20683268
- [Background] Zelenetz AD, Abramson JS, Advani RH, Andreadis CB, Byrd JC, Czuczman MS, Fayad L, Forero A, Glenn MJ, Gockerman JP, Gordon LI, Harris NL, Hoppe RT, Horwitz SM, Kaminski MS, Kim YH, Lacasce AS, Mughal TI, Nademanee A, Porcu P, Press O, Prosnitz L, Reddy N, Smith MR, Sokol L, Swinnen L, Vose JM, Wierda WG, Yahalom J, Yunus F. NCCN Clinical Practice Guidelines in Oncology: non-Hodgkin's lymphomas. J Natl Compr Canc Netw. 2010 Mar;8(3):288-334. doi: 10.6004/jnccn.2010.0021. No abstract available. PMID 20202462